CLINICAL TRIAL: NCT00372645
Title: Effects Of A Mixed Diet Intervention Versus Folic Acid Supplementation And Metafolin® Supplementation On Folate Status And Cardiovascular Disease Risk Factors In Healthy Adults
Brief Title: Increasing Folate Status of a General Population(FOLSUPP STUDY)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Food Standards Agency, United Kingdom (Other Government); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: IFR001/2005; NORFOLK LREC 05/Q0101/51; FSA GRANT NUMBER N05057; IFR PROJECT NUMBER 51943F
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Healthy
MeSH Terms: interventions — Folic Acid; levomefolate calcium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diet (Experimental): 200 µg folate per day from folate-rich foods
  Interventions: Other: Folate rich foods
- Folic acid supplement (Experimental): 200 µg folate per day from supplemental folic acid
  Interventions: Dietary Supplement: Folic acid (supplement)
- Metfolin supplement (Experimental): 200 µg folate per day from supplemental Metafolin®
  Interventions: Dietary Supplement: Metafolin (supplement)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Folic acid (supplement) — 200 µg folate per day from supplemental folic acid
  Arms: Folic acid supplement
Dietary Supplement: Metafolin (supplement) — 200 µg folate per day from supplemental Metafolin®
  Arms: Metfolin supplement
Drug: Placebo — Placebo
  Arms: Placebo
Other: Folate rich foods — 200 µg folate per day from folate-rich foods
  Arms: Diet

SUMMARY:
The aim of this study is to determine the best source of folate to raise the folate status of a general population over a 16 week intervention period.

DETAILED DESCRIPTION:
This study is designed to assess whether increasing the consumption of natural food folates from a mixed diet is as effective as supplemental folic acid or supplemental natural folate in raising folate status, reducing biomarkers of cardio vascular disease (CVD) risk, and improving vascular function. Randomised placebo-controlled parallel studies will be undertaken in groups of individuals in Norwich and Sheffield. There will be four treatment arms: a) 200 µg folate per day from folate-rich foods, b) 200 µg folate per day from supplemental folic acid, c) 200 µg folate per day from supplemental Metafolin® (6S 5-methyltetrahydrofolic acid) and d) a placebo group. Results from the two centres will be combined, thus ensuring a wide population is covered. Folate status, biomarkers of CVD risk and vascular function (pulse wave velocity) will be measured before and following the intervention period of 16 weeks, together with possible confounders (such as vitamins B2 & B12 status, and MTHFR genotype). 7-Day weighed intakes will be used to measure habitual B-vitamin intake during baseline and intervention, to determine changes in folate intake and assist compliance. Additionally, folate content of selected folate-rich foods will be determined for each volunteer. The results will aid the Food Standards Agency (FSA) in formulating public health policy related to improving folate status and reducing CVD risk.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-65 years
* Smokers and non-smokers

Exclusion Criteria:

* Pregnant or has been pregnant within the last 12 months
* Breastfeeding
* Has donated or intends to donate blood within 16 weeks of the first or last study samples
* Fails standard clinical screening of blood and urine for human studies at the Institute of Food Reseach
* BMI above 18 or below 40
* Receiving vascular disease or anti-hypertensive drugs
* Those with diabetes
* Regularly consuming dietary supplements containing B-vitamins and/or folic acid.

[As the capsules are prepared from gelatin, true vegetarians may not wish to participate]

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-05; Primary Completion 2008-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Folate status | Baseline and 16 weeks
Homocysteine status | Baseline and 16 weeks

SECONDARY OUTCOMES:
Cardio vascular disease markers | Baseline and 16 weeks
Inflammatory markers | Baseline and 16 weeks
Pulse wave velocity | Baseline and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Flingas, BSc, Principal Investigator — Quadram Institute Bioscience; Hilary Powers, BSc PhD, Principal Investigator — University of Sheffield
Locations (2):
- United Kingdom (2):
  - Institute of Food Research, Norwich, Norfolk
  - University of Sheffield, Sheffield, Yorkshire

REFERENCES:
- See also: Institute of Food Research home page — http://www.ifr.ac.uk